CLINICAL TRIAL: NCT00923611
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Grouped, Clinical Study to Evaluate the Antihypertensive Efficacy and Tolerability and to Determine the Adequate Antihypertensive Dosage of Fimasartan(BR-A-657-K) in Patients With Mild to Moderate Essential Hypertension
Brief Title: Antihypertensive Efficacy and Tolerability and Determine the Adequate Antihypertensive Dosage of Fimasartan in Mild to Moderate Essential Hypertension Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Collaborators: Seoul National University Hospital (Other); Samsung Medical Center (Other); Asan Medical Center (Other); Seoul National University Bundang Hospital (Other); The Catholic University of Korea (Other); Severance Hospital (Other); Yonsei University (Other); Cheil General Hospital and Women's Healthcare Center (Other)
Responsible Party: Choi, Director, Boryung Pharm Co., Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A-657-BR-CT-202
Record Dates: First submitted 2009-06-16; First posted 2009-06-18 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2009-06

CONDITIONS: Hypertension
Keywords: Hypertension; Fimasartan
MeSH Terms: conditions — Hypertension | interventions — fimasartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): 3 tablets of placebo will be taken 30minutes after breakfast for 8 weeks
  Interventions: Drug: Fimasartan
- Fimasartan 20mg (Active Comparator): 2 tablets of placebo and 1 tablets of fimasartan 20mg will be taken 30minutes after breakfast for 8 weeks
  Interventions: Drug: Fimasartan
- Fimasartan 60mg (Active Comparator): 3 tablets of fimasartan 20mg will be taken 30minutes after breakfast for 8 weeks
  Interventions: Drug: Fimasartan
- Fimasartan 120mg (Active Comparator): 3 tablets of fimasartan 40mg will be taken 30minutes after breakfast
  Interventions: Drug: Fimasartan
- Fimasartan 240mg (Active Comparator): 3 tablets of fimasartan 80mg will be taken 30minutes after breakfast for 8 weeks
  Interventions: Drug: Fimasartan

INTERVENTIONS:
Drug: Fimasartan

SUMMARY:
The purpose of this study is to evaluate the antihypertensive efficacy and tolerability of 8 week treatment with Fimasartan (BR-A-657-K) 20, 60, 120, 240 mg and placebo in patients with mild to moderate essential hypertension and to determine the adequate antihypertensive dosage for later clinical study.

DETAILED DESCRIPTION:
Fimasartan (BR-A-657-K), a selective blocker of AT1 receptor subtype, showed the rapid and potent antihypertensive effect in many hypertensive models. Phase I study, Fimasartan (BR-A-657-K) 20mg ~ 480mg single dosing with healthy subjects, demonstrated that the Fimasartan (BR-A-657-K) was very safe and well tolerated. Another phase I study, Fimasartan (BR-A-657-K) 120mg and 360mg dosing for 7 days, also showed that Fimasartan (BR-A-657-K) was safe and tolerable though one temporal adverse event was observed in high dose.

A randomized, double-blind, placebo-controlled, parallel grouped, clinical study will be conducted to evaluate the antihypertensive efficacy and tolerability and to determine adequate antihypertensive dosage of Fimasartan(BR-A-657-K) in patients with mild to moderate essential hypertension.

Approximately 182 patients will be enrolled over 12 months in 8 centers nationwide.

After 2 weeks of placebo run-in period, all subjects will be randomized into one of the following 5 groups. Subjects will take test/control drug for 8 weeks of treatment period. If subjects take any antihypertensive medications before screening, the subjects will have 1 week of wash-out period.

Group I : Placebo, Group II : Fimasartan 20 mg, Group III: Fimasartan 60 mg, Group IV : Fimasartan 120 mg, Group V : Fimasartan 240 mg,

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate essential hypertension : sitting diastolic blood pressure measured at Screening and Baseline(Day1) are 95~114 mmHg inclusive and the difference between sitting diastolic blood pressures measured at Day -14 and Baseline(Day1) is under 7mmHg.
* Subjects who agree to participate in this sudy and give written informed consent
* Subjects considered to understand the study, be cooperative, and able to be followed-up until the end of the study

Exclusion Criteria:

* The sitting DBP is less than 94mmHg or more than 115mmHg or severe hypertensive patient with sitting systolic blood pressure over 200mmHg
* Patients with secondary hypertension
* Patients with severe renal(Creatinine more 1.5 times than upper limit of normal), gastrointestinal, hematological or hepatic(AST, ALT more 2 twice more than upper limit of normal)disease etc. which might affect absorption, disposition, metabolism or excretion of the drug
* Patients with postural hypotension
* Patients with sever insulin dependent diabetes mellitus or uncontrolled diabetes mellitus(HbA1c>9%, regimen change of oral hypoglycemic agents within 3 months, treated insulin before screening)
* Patients with a history of myocardial infarction, severe coronary artery disease or clinically significant heart failure or valvular defect in last 6 months
* Patients with consumptive disease, autoimmune disease, connective tissue disease
* Patients with a history of type B or C hepatitis
* Patients with HIV or hepatitis
* Patients with clinically significant laboratory abnormality
* Patients receiving any drugs known to affect blood pressure or medical treatments that can influence the blood pressure
* Patients with allergy or contraindication to any angiotensin II receptor antagonists
* Female of childbearing potential who does not undergo hysterectomy or is not post-menopausal
* Patients judged to have a history of alcohol or drug abuse by the investigator
* Patients with average weight > +35% or <-15% in Modified Metropolitan Life Insurance table
* Patients participated other clinical trial 3 months before Screening
* Patients judged to be inappropriate for this study by the investigator with other reasons

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
change from baseline to end of 8 week treatment in sitting diastolic blood pressure | 8 week from baseline

SECONDARY OUTCOMES:
change from baseline to end of 2,4 week treatment in sitting diastolic blood pressure | 2, 4 week from baseline
change from baseline to end of 2,4,8 week treatment in sitting systolic blood pressure | 2,4,8 week from baseline
responders after end of 8 week treatment(portion of DBP<90mmHg or the difference from baseline and end of 8 week treatment>10mmHg | 8 week from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Hee Oh, Professor, Study Chair — Seoul National University Hospital; Jae-Joong Kim, Professor, Principal Investigator — Asan Medical Center; Eun-Suk Jeon, Professor, Principal Investigator — Samsung Medical Center; Dong-Ju Choi, Professor, Principal Investigator — Seoul National University Bundang Hospital; Ki-Bae Seong, Professor, Principal Investigator — Kangnam ST.Mary's Hospital; Jong-Won Ha, Professor, Principal Investigator — Severance Hospital; Se-Joong Lim, Professor, Principal Investigator — Yonsei University; Jeong-Bae Park, Professor, Principal Investigator — Cheil General Hospital and Women's Healthcare Center
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee H, Yang HM, Lee HY, Kim JJ, Choi DJ, Seung KB, Jeon ES, Ha JW, Rim SJ, Park JB, Shin JH, Oh BH. Efficacy and tolerability of once-daily oral fimasartan 20 to 240 mg/d in Korean Patients with hypertension: findings from Two Phase II, randomized, double-blind, placebo-controlled studies. Clin Ther. 2012 Jun;34(6):1273-89. doi: 10.1016/j.clinthera.2012.04.021. Epub 2012 May 17. PMID 22608107